CLINICAL TRIAL: NCT00000278
Title: Disulfiram for Cocaine-Alcohol Abuse
Brief Title: Disulfiram for Cocaine-Alcohol Abuse - 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-09250-3; P50DA009250 (NIH); P50-09250-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Alcohol-Related Disorders; Cocaine-Related Disorders
Keywords: Cocaine-Related Disorders
MeSH Terms: conditions — Alcohol-Related Disorders; Cocaine-Related Disorders | interventions — Disulfiram

INTERVENTIONS:
Drug: Disulfiram

SUMMARY:
The purpose of this study is to evaluate disulfiram for cocaine-alcohol abuse.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1994-09; Primary Completion 1999-08 (Actual); Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Side effects
Cocaine effects

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kosten, M.D., Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, New Haven, Connecticut, United States

REFERENCES:
- [Background] Biol Psy. 37: 560-563, 1995. NIDA Research Monograph, 174:138, 1997. Ther Drug Monograph, 18:460-464, 1996.
- [Derived] Traccis F, Minozzi S, Trogu E, Vacca R, Vecchi S, Pani PP, Agabio R. Disulfiram for the treatment of cocaine dependence. Cochrane Database Syst Rev. 2024 Jan 5;1(1):CD007024. doi: 10.1002/14651858.CD007024.pub3. PMID 38180268